CLINICAL TRIAL: NCT05328856
Title: An Randomised Controlled Trial on the Effects of Vital Shower (Hansgrohe) on Quality of Life, Immune Function, Cardiovascular Regulation and Well-being
Brief Title: Effects of Vital Shower on Quality of Life, Immune Function, Cardiovascular Regulation and Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VD
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: General Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vital shower (Active Comparator): Participants receive a prototype/shower head from Hansgrohe and training including a handout. After installation, participants are asked to shower daily for four weeks according to a predefined shower protocol.
  Interventions: Device: Hansgrohe prototype/shower head
- Regular shower (No Intervention): Participants are advised not to change their showering behaviour; at the end of the study, the participants receive an offer of a shower head for free.

INTERVENTIONS:
Device: Hansgrohe prototype/shower head — Start of the shower with warm comfort temperature and usual body cleansing. Then the Vital shower is carried out for a total of 3-5 minutes, followed optionally by another warm shower with 30 seconds or direct transition to a classic cold shower for 30- 60 seconds
  Arms: Vital shower

SUMMARY:
The aim of this exploratory randomized controlled clinical study is to evaluate the health-promoting effects of Kneipp hydrotherapy, in the form of the Vital Shower in a four-week daily application.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients between 18 and 70 years of age

Exclusion Criteria:

* Bad general condition
* Serious acute or chronic comorbidity
* Pregnancy and breast feeding period/ in the next 6 months
* Participation in a clinical trial within the last 3 months before enrollment
* Simultaneous participation in another clinical trial
* Raynaud's disease or cold agglutinin disease
* Severe mental illness
* Insufficiently treated dermatological diseases (e.g. neurodermatitis, psoriasis)
* Non-compatible sanitary shower or bath devices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunological laboratory | Change from Baseline and after 4 weeks
  T-Cells (CD3), B-Cells (CD19), Natural Killer Cells (CD16), T-helper cells (CD4), cytotoxic T-cells (CD8), CD4/CD8 ratio, interleukin 4, interferon gamma
Blood pressure at rest (systolic and diastolic) | Change from Baseline and after 4 weeks
Hospital Anxiety and Depression Scale (HADS-D) | Change from HADS-D Baseline, after 4 weeks and 12 weeks
  Change
Self-Efficacy Scale (ASKU) | Change from ASKU Baseline, after 4 weeks and 12 weeks
  Change
WHO-Five Well-Being Index (WHO-5) | Change from WHO-5 Baseline, after 4 weeks and 12 weeks
  Change
Perceived Stress Scale (PSS-10) | Change from PSS-10 Baseline, after 4 weeks and 12 weeks
  Change
Flourishing Scale (FS-D) | Change from FS-D Baseline, after 4 weeks and 12 weeks
  Change
Insomnia Severity Index (ISI-D) | Change from ISI-D Baseline, after 4 weeks and 12 weeks
  Change
Short Form (SF-36) | Change from SF-36 Baseline, after 4 weeks and 12 weeks
  Change
Von Zerssen somatic complaint list (B-LR and B-LR') | Change from B-LR and B-LR' Baseline, after 4 weeks and 12 weeks
  Change
Heart rate variability | Change from Baseline and after 4 weeks
  Change

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, State of Berlin, Germany